CLINICAL TRIAL: NCT01026688
Title: Evaluation of a Toolkit to Improve Cardiovascular Disease Screening and Treatment for People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Shah-1
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes Mellitus; Cardiovascular Disease
Keywords: Pragmatic randomized controlled trial; Cardiovascular risk reduction; Knowledge translation; Clinical practice guidelines
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Toolkit
- Control (Other)
  Interventions: Other: Control

INTERVENTIONS:
Other: Toolkit — Cardiovascular Disease Toolkit mailed by the Canadian Diabetes Association to family physicians, accompanying the Spring/Summer 2009 edition of the quarterly newsletter, Canadian Diabetes. (Mailed in June 2009.) The Toolkit includes a summary of selected sections of the practice guidelines targeted towards primary care physicians; a synopsis of the key messages pertaining to cardiovascular disease risk; a laminated card with a simplified algorithm for cardiovascular risk assessment and treatment; and a pad of tear-off sheets for patients with a cardiovascular risk self-assessment tool.
  Arms: Intervention
Other: Control — The Spring/Summer 2009 issue of the quarterly newsletter, Canadian Diabetes, mailed on its own. The Cardiovascular Toolkit was mailed to Control arm physicians with the May 2010 issue of the newsletter.
  Arms: Control

SUMMARY:
Diabetes is a common and serious chronic disease. However, there is a large gap between the level of care that people should receive (based on research and guidelines) and the level of care they actually receive. With the release of their 2008 Clinical Practice Guidelines, the Canadian Diabetes Association has a strategy to improve heart disease screening and treatment for people with diabetes. This study will evaluate whether the strategy works. The focus of the strategy was to give all family physicians in Canada a Toolkit in June 2009 to help them delivery better care for their diabetic patients. In Ontario, only half of doctors received this Toolkit. We will compare the quality of care received by diabetic patients whose doctors received this Toolkit versus those who doctors did not.

DETAILED DESCRIPTION:
A cardiovascular disease Toolkit was developed by the Canadian Diabetes Association and mailed to family physician with the Spring/Summer 2009 edition of the newsletter, Canadian Diabetes. The Toolkit was packaged in a brightly-coloured box with Canadian Diabetes Association branding, and contained: 1) an introductory letter from the Chair of the practice guidelines' Dissemination and Implementation Committee; 2) an eight page summary of selected sections of the practice guidelines targeted towards primary care physicians; 3) a four page synopsis of the key guideline elements pertaining to cardiovascular disease risk; 4) a small double-sided laminated card with a simplified algorithm for cardiovascular risk assessment, vascular protection strategies and screening for cardiovascular disease; and 5) a pad of tear-off sheets for patients with a cardiovascular risk self-assessment tool and a list of recommended risk reduction strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed diabetes
* Seen in the office of a participating family physician at least once between July 2009 and April 2010
* At high risk for cardiovascular events:

  * Previous cardiovascular disease (including AMI, angina, stroke, TIA, claudication); or
  * Men aged >= 45 years, women aged >= 50 years; or
  * Men aged < 45 years, women aged < 50 years with at least one of the following:

    1. Macrovascular disease (silent myocardial infarction, or evidence of peripheral arterial, carotid or cerebrovascular disease)
    2. Microvascular disease (nephropathy or retinopathy)
    3. Family history of premature coronary or cerebrovascular disease in a first-degree relative
    4. Duration of diabetes > 15 years with age > 30 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1592 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Patient is receiving a statin | July 2009 to April 2010

SECONDARY OUTCOMES:
Patient is receiving an angiotensin-converting enzyme inhibitor or angiotensin receptor blocker | July 2009 to April 2010
A1c level | Last observation between July 2009 and April 2010
Blood pressure level | Last observation between July 2009 and April 2010
LDL-cholesterol level | Last observation between July 2009 and April 2010
Total- to HDL-cholesterol ratio | Last observation between July 2009 and April 2010
Body mass index | Last observation between July 2009 and April 2010
Waist circumference | Last observation between July 2009 and April 2010
Change in treatment recommended following an A1c level above 0.070 | At the next patient visit after the abnormal measurement
Change in treatment recommended following a systolic blood pressure above 130 or a diastolic blood pressure above 80 | At the patient visit of the abnormal measurement
Change in treatment recommended following an LDL-cholesterol level above 2.0 mmol/L | At the next patient visit after the abnormal measurement

CONTACTS AND LOCATIONS:
Overall Officials: Baiju R Shah, MD PhD, Principal Investigator — Institute for Clinical Evaluative Sciences
Locations (1):
- Institute for Clinical Evaluative Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Background] Shah BR, Bhattacharyya O, Yu CH, Mamdani MM, Parsons JA, Straus SE, Zwarenstein M. Effect of an educational toolkit on quality of care: a pragmatic cluster randomized trial. PLoS Med. 2014 Feb 4;11(2):e1001588. doi: 10.1371/journal.pmed.1001588. eCollection 2014 Feb. PMID 24505216
- [Derived] Shah BR, Bhattacharyya O, Yu C, Mamdani M, Parsons JA, Straus SE, Zwarenstein M. Evaluation of a toolkit to improve cardiovascular disease screening and treatment for people with type 2 diabetes: protocol for a cluster-randomized pragmatic trial. Trials. 2010 Apr 23;11:44. doi: 10.1186/1745-6215-11-44. PMID 20416080